CLINICAL TRIAL: NCT04490122
Title: Impact of Mode of Anesthesia on Ischemia Modified Albumin (Abiomarker of Oxidative Stress) and Outcome in Patients With Traumatic Brain Injury Undergoing Emergency Craniotomy
Brief Title: Impact of Mode of Anesthesia on Ischemia Modified Albumin in Patients With Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Abd-elrahman hassan abd -elaziz (Other)
Responsible Party: Sponsor-Investigator, Abd-elrahman hassan abd -elaziz, Minia University Hospital, Minia University
Organization: Minia University (Other)
Other Study IDs: 374
Record Dates: First submitted 2020-02-23; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-02

CONDITIONS: Oxidative Stress
Keywords: Ischemia modified albumin; oxidative stress; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhalational: will receive inhalational anesthesia
- Total intravenous: will receive total intravenous anesthesia with propofol infusion(100-150 mcg/kg/min) and dexmedetomedine 0.3mcg/kg/h.

SUMMARY:
In the current study the investigators intend to evaluate the mode of anesthesia on ischemia modified albumin and outcome in patients with traumatic brain injury undergoing emergency craniotomy

DETAILED DESCRIPTION:
After obtaining Institutional Ethical Committee approval and written informed consent from legally acceptable representative relatives, patients with traumatic brain injury, aged from 18- 60 years old, ASA from (I-III), GCS more than 8 undergoing emergency craniotomy surgery will be selected for this prospective randomized Study.

The anesthesia will be induced with 2mcg/kg fentanyl and 2 mg/kg propofol. Muscle relaxation will be achieved with 0.5 mg/kg atracurium.

Anesthesia will be maintained with:

* Group I, isoflurane (mac<1) mixed with oxygen 40% and fentanyl 1mcg/kg hourly.
* Group PD, propofol infusion(100-150mcg/kg/min) and dexmedetomedine 0.3mcg/kg /h.

Parameters will be assessed Preoperative period

* Ischemia modified albumin level from venous sample.
* Basal Systolic blood pressure, diastolic blood pressure. Mean arterial blood pressure, oxygen saturation, heart rate.
* GCS. Intraoperative period
* Systolic blood pressure, diastolic blood pressure. Mean arterial blood pressure, oxygen saturation, heart rate after intubation, 5,15,30,60,90min and after extubation.
* Need for resuscitation with vasoactive drugs.
* Brain relaxation score at dural opening and closure.
* ICP
* Intraoperative blood loss.
* Amount of fluid and blood transfusion. Postoperative period
* Ischemia modified albumin immediately postoperatively, after 6h and after 24 hours.
* Type of surgery.
* Duration of surgery.
* Extubation time.
* Recovery scores (Ramsay sedation score and modified Alderte score).
* GCS immediately postoperatively, after 6h, after 24h and after 48 hours.
* Total analgesic requirement during the first 24 hours.
* Need for ICU admission.
* Length of ICU stay.
* Complications.
* 28 day mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old of both sex .
2. Isolated traumatic brain injury undergoing emergency craniotomy.
3. G.C.S more than 8.
4. ASA grade (I-III).

Exclusion Criteria:

1. Non traumatic brain injury.
2. Poly trauma patient.
3. Coagulation disorder.
4. Drug( alcohol, opiods, tranquilizers) addiction.
5. Liver and kidney dysfunction.
6. Severe diseases such as severe hypertension, cardiovascular disease, malignant tumor, autoimmune disease, mental disorders.
7. Diabetes mellitus with poor blood glucose control.
8. Previous drug allergy.
9. Currently lactating.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with traumatic brain injury, aged from 18- 60 years old, ASA from (I-III), GCS more than 8 undergoing emergency craniotomy surgery
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2020-07-23 (Estimated); Primary Completion 2021-07-28 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
ischemia modified albumin | change from preoperative level of ischemia modified albumin at the first 24 hours postoperatively
  Plasma Level of ischemia modified albumin
Glascow Coma Scale | change from preoperative Glascow Coma Scale score at the first 24 hours postoperatively
  Glascow Coma Scale records the state of a person's consciousness. it gives a person's score between 3 (indicating deep unconsciousness) and 15 (indicating fully consciousness)

SECONDARY OUTCOMES:
Intraoperative blood pressure. | preoperatively, immediatly after intubation,after 5 minutes,afer 15 minutes,after 30 minutes,after 60 minutes,after 90 minutes and immediatly after extubation.
  Intraoperative haemodynamics (Systolic blood pressure in millimeter mercury, diastolic blood pressure in millimeter mercury. Mean arterial blood pressure in millimeter mercury.
Intraoperative heart rate | preoperatively, immediatly after intubation,after 5 minutes,afer 15 minutes,after 30 minutes,after 60 minutes,after 90 minutes and immediatly after extubation.
  Intraoperative heart rate per minute
I.C.U admission | up to 28 days
  intensive care unit admission
I.C.U stay. | up to 28 days
  Length of stay in intensive care unit
Incidence of any complication. | up to 28 days
  Incidence of any complication (nausea, vomiting, convulsion and reopening).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K Mohamed, professor, Principal Investigator — Minia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Decompressive craniectomy and traumatic brain injury: a review. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4771225/
- See also: Comparison of total intravenous anesthesia vs. inhalational anesthesia on brain relaxation, intracranial pressure, and hemodynamics in patients with acute subdural hematoma undergoing emergency craniotomy: a randomized control trial — https://www.ncbi.nlm.nih.gov/pubmed/31664468
- See also: The comparison of the effects of sevoflurane inhalation anesthesia and intravenous propofol anesthesia on oxidative stress in one lung ventilation. — https://www.ncbi.nlm.nih.gov/pubmed/24527444